CLINICAL TRIAL: NCT06973239
Title: Evaluation of the Safety and Performance of the Neocement® Inject P: A Prospective Observational Study in Orthopaedic Area
Brief Title: Evaluation of the Safety and Performance of the Neocement® Inject P
Status: Recruiting | Type: Observational
Sponsor: Bioceramed (Industry)
Collaborators: Local Health Unit Barcelos/Esposende, Public Health Unit (Other Government)
Responsible Party: Sponsor
Other Study IDs: NeocementInject01
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Bone Defects; Orthopaedic Surgery (30 Minutes or Longer)
Keywords: Neocement® Inject P; prospective observational clinical study; medical device; performance and safety; bone defects; real-world clinical data; post-market; calcium phosphates; synthetic bone substitute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to collect real-world clinical data to gather information on the performance and safety of the Neocement® Inject P when used according to its intended purpose and current clinical applications. The results of the clinical study will serve as clinical evidence for the device's clinical evaluation, targeting submission to the new Medical Device Regulation (EU) 2017/745.

DETAILED DESCRIPTION:
Neocement® Inject P represents a breakthrough in orthopaedic biomaterials, meticulously engineered to enhance bone repair and regeneration. This synthetic bone substitute combines tetracalcium phosphate and beta-tricalcium phosphate within its P-system architecture, augmented by chitosan and an aqueous solution enriched with citric acid and glucose.

Neocement® Inject P is indicated for filling bony voids or gaps of the skeletal system that are not intrinsic to the stability of the bony structure. The device may be used for filling surgically created bone defects or osseous defects created from traumatic injury to the bone.

To achieve its intended purpose, Neocement® Inject P will be placed in contact with bone tissue and surrounding tissues by surgically invasive techniques in operating rooms. More than one unit of Neocement® Inject P can be used for filling bony voids or gaps of the skeletal system, depending on the lesion.

Neocement® Inject P is a class III medical device. This advanced biomaterial offers a reliable solution for addressing bone fractures and loss, demonstrating significant potential in enhancing patient outcomes through accelerated and durable bone regeneration. Neocement® Inject P is expected to be partially or totally resorbed, from the clinical available data, the expected effect can be predicted to occur after 6 months.

This observational post-market study will collect data relating to standard practice procedures, therefore there are no additional risks or direct benefits associated with participating in this registry for the patient.

This study based on observations of clinical practice aims to collect clinical data to keep up to date the information on the performance and safety of the medical device when used in accordance with its intended use and current clinical applications. The results of the clinical study shall be used as clinical evidence for clinical evaluation of the device aiming submission to the new Medical Device Regulation (EU) 2017/745.

The post-market study is meant to identify and analyse emerging risks, ensure the continued acceptability of the benefit/risk ratio and also identify possible systematic misuse or unauthorized use of the medical device. This protocol does not include any planned new uses, new populations, new materials or design changes.

The results from the prospective observational post-market study will provide an evidence base for assessing the device's performance and safety after its market launch. Detecting real discrepancies in clinical performance between of the medical device early on can offer valuable opportunities to improve device design. This complements the data collected during the pre-market phases, thus improving patient selection. Active surveillance of the safety of medical devices, achieved through the continuous monitoring of vast sources of clinical data, is a priority in the field of medical devices, a requirement of MDR regulation No. 2017/745. This approach is crucial to achieving the objectives set, guaranteeing the safety and performance of the devices in circulation.

Patients will be followed as per local standard medical practices of the centre for 1 year.

Clinical data will be collected at 4 points in time: Visit 1 (6 weeks ± 2 weeks - enrolment), Visit 2 (3 months ±3 weeks), Visit 3 (6 months ±3 weeks) and if necessary, a Visit 4 (12 months ±30 days).

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females (age > 18 years old);
* Patients with bone defect treatment who meet predefined criteria in Instructions For Use (IFU) of Neocement® Inject P;
* Patients who are able to sign an informed consent form (for data collection)
* Patients with bone defects, which may be surgically created or result from traumatic injury to the bone;
* Patients with bone skeletal defects that are not intrinsic to the stability of the bone structure or with a site that can be stabilized;

Exclusion Criteria:

* Patients who are unable to understand consent and the objectives of the study;
* Signs of local or systemic acute/ active or chronic infections;
* Metabolic affections;
* Severe degenerative diseases, conditions in which general bone grafting is not advisable;
* Implementation sites that allow product migration;
* Conditions which require structural support in the skeletal system;
* Conditions where the implantation site is unstable and not rigidly fixated;
* Sensibility to the implantable materials;
* Known hypersensitivity to the implant material.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The clinical study population consists of adult patients (aged > 18 years old) undergoing orthopaedic surgery to treat bone defects. It is expected that clinical data will be collected from 80 patients implanted with the Neocement® Inject P product.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Performance Endpoint | 6 weeks; 3 months; 6 months and 12 months (if necessary)
  Bone consolidation on the surgery site (discrete variable: Yes or No), assessed by X-ray or CT scan.
Safety Endpoint | 6 weeks; 3 months; 6 months and 12 months (if necessary)
  The assessment of Adverse Events and Device deficiencies at least possibly related to Neocement® Inject P during the follow-up period of patients.

SECONDARY OUTCOMES:
Quality of life measured through the Short Form Health Survey (SF-36) Questionnaire | 6 weeks after surgery; 6 months
  Quality of life will be assessed during the patients' follow-up period. Patients will complete the SF-36 questionnaire to assess quality of life and to measure the Health Status during recovery.
  The SF-36 (Short Form Health Survey) is a questionnaire widely used to assess health-related quality of life. Composed of 36 questions, it covers eight main dimensions: physical functioning, limitations due to physical aspects, pain, general health status, vitality, social functioning, limitations due to emotional aspects and mental health. The score in each dimension allows a comprehensive analysis of the patient's perception of their physical and mental well-being, making it a valuable tool both in clinical research and in medical practice for monitoring the health of individuals and populations.
Surgeon's Satisfaction survey on the medical device and Technical Success; | 6 weeks after surgery
  To evaluate the Technical Success rate, defined as the successful delivery of the bone substitute into the target defect without any malfunction of the delivery device or the bone substitute itself, and to collect usability feedback on the device during the surgical procedure through a Satisfaction survey.
  Information on the surgeon's satisfaction with the device under study should be collected post-operatively through a general questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Unidade Local de Saúde Esposende/Barcelos, Barcelos, Portugal

IPD SHARING:
Plan to Share IPD: No